CLINICAL TRIAL: NCT00270751
Title: Comparison of Pleural Abrasion Plus Minocycline Pleurodesis Versus Apical Pleurectomy After Thoracoscopic Bullectomy for High Recurrent Risk Patients With Primary Spontaneous Pneumothorax: A Prospective Randomized Trial.
Brief Title: Pleural Abrasion Plus Minocycline Versus Apical Pleurectomy for Primary Spontaneous Pneumothorax
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31MD02
Record Dates: First submitted 2005-12-26; First posted 2005-12-28 (Estimated); Last update posted 2006-08-07 (Estimated); Status verified 2006-08

CONDITIONS: Pneumothorax
Keywords: Video-Assisted Thoracoscopic Surgery; Spontaneous pneumothorax; Pleurectomy; Pleural abrasion; Minocycline
MeSH Terms: conditions — Pneumothorax; cyclopia sequence

INTERVENTIONS:
Procedure: 1 apical pleurectomy
Procedure: 2 pleural abrasion + minocycline pleurodesis

SUMMARY:
Optimal surgical management of primary spontaneous pneumothorax has been a matter of devate, especially regarding the method of pleurodesis. Previous studies have shown that thoracoscopic apical pleurectomy is a reliable method with a very low incidence of recurrence. However, this procedure is more technical demanding and time consuming through thoracoscopy. In addition, a more extensive pleural injury may cause impaired pulmonary function and a higher risk of perioperative complication such as hemothorax. In our previous studies, we have shown that thoracoscopic pleural abrasion with minocycline instillation is an easy and convinent method of pleurodesis which decreases the rate of recurrence without affecting pulmonary function. In this study, we hypothesized that pleural abrasion with minocycline instillation is as effective as apical pleurectomy in preventing pneumothorax recurrence while the short-term and long-term complications are less.

DETAILED DESCRIPTION:
Optimal surgical management of primary spontaneous pneumothorax has been a matter of devate, especially regarding the method of pleurodesis. Previous studies have shown that thoracoscopic apical pleurectomy is a reliable method with a very low incidence of recurrence. However, this procedure is more technical demanding and time consuming through thoracoscopy. In addition, a more extensive pleural injury may cause impaired pulmonary function and a higher risk of perioperative complication such as hemothorax. In our previous studies, we have shown that thoracoscopic pleural abrasion with minocycline instillation is an easy and convinent method of pleurodesis which decreases the rate of recurrence without affecting pulmonary function. In this study, we hypothesized that pleural abrasion with minocycline instillation is as effective as apical pleurectomy in preventing pneumothorax recurrence while the short-term and long-term complications are less.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 50 years old Undergoing thoracoscopic bullectomy Had multiple blebs or no identified blebs during the operation

Exclusion Criteria:

* With underlying pulmonary disease With major systemic disease or acute infection Underwent ipsilateral operation previously Bleb number = 1 or 2

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2005-04; Study Completion 2009-05

PRIMARY OUTCOMES:
Recurrence rate of pneumothorax after thoracoscopic operation.

SECONDARY OUTCOMES:
The short-term results (Pain level, chest tube duration, hospital stay, etc)
Complication rate
Long-term results: residual pain
Long-term pulmonary function test

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, MD, PhD, Study Chair — Department of Surgery, National Taiwan University Hospital, Taiwan; Jin-Shing Chen, MD, PhD, Study Director — Department of Surgery, National Taiwan University Hospital, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Chen JS, Hsu HH, Chen RJ, Kuo SW, Huang PM, Tsai PR, Lee JM, Lee YC. Additional minocycline pleurodesis after thoracoscopic surgery for primary spontaneous pneumothorax. Am J Respir Crit Care Med. 2006 Mar 1;173(5):548-54. doi: 10.1164/rccm.200509-1414OC. Epub 2005 Dec 15. PMID 16357330
- [Background] Chen JS, Hsu HH, Kuo SW, Tsai PR, Chen RJ, Lee JM, Lee YC. Effects of additional minocycline pleurodesis after thoracoscopic procedures for primary spontaneous pneumothorax. Chest. 2004 Jan;125(1):50-5. doi: 10.1378/chest.125.1.50. PMID 14718420
- [Derived] Chen JS, Hsu HH, Huang PM, Kuo SW, Lin MW, Chang CC, Lee JM. Thoracoscopic pleurodesis for primary spontaneous pneumothorax with high recurrence risk: a prospective randomized trial. Ann Surg. 2012 Mar;255(3):440-5. doi: 10.1097/SLA.0b013e31824723f4. PMID 22323011